CLINICAL TRIAL: NCT02007369
Title: Effectiveness of Using Social Networking Service to Prevent Smoking Relapse Among Self-reported Quitters: A Pilot Randomized Control Trial
Brief Title: Relapse Prevention Through Social Networking Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Tung Wah Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TWRP2013
Record Dates: First submitted 2013-11-28; First posted 2013-12-10 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- WhatsApp (Experimental): Provide peer support and deliver relapse prevention messages through WhatsApp for 8 weeks and telephone follow ups
  Interventions: Behavioral: WhatsApp
- Facebook (Experimental): Provide peer support and deliver relapse prevention messages through Facebook for 8 weeks and telephone follow ups
  Interventions: Behavioral: Facebook
- Control (No Intervention): Telephone follow ups and received a self-help book only

INTERVENTIONS:
Behavioral: WhatsApp — Intervention arm with relapse prevention intervention in the social group via the social networking service WhatsApp and the duration of the intervention will be 8 weeks.
  Arms: WhatsApp
Behavioral: Facebook — Another intervention arm with the same intervention content, but the platform for the participants to share and receive quitting advice is Facebook and the duration of the intervention will be 8 weeks.
  Arms: Facebook

SUMMARY:
According to the Census & Statistics Department, there are still 659,300 daily smokers (11.1%) in Hong Kong. Smoking is addictive, and it is difficult for some motivated smokers to quit without assistance. About 33.2% daily smokers in Hong Kong had tried quitting but they could not maintain abstinence. Relapse prevention is aimed at providing interventions to prevent relapse after starting the abstinence status. This pilot single-blind randomized controlled trial (proof of concept study) will test the effectiveness of social networking services for relapse prevention. The study will first recruit 6 quitters and 6 relapsers for a qualitative interview for the design of intervention. Then, the pilot-RCT trial will recruit 120 participants who have recently quitted smoking, and they will be randomly allocated to 2 intervention groups and one control group. The 2 intervention groups will be arranged to join a WhatsApp or Facebook group for receiving quitting advices from the group moderators and sharing quitting experience with other participants. All participants will receive a self-help booklet of relapse prevention, and will be followed up at 6 weeks, 3 months and 6 months. The primary outcome is the self-report relapse rate (Relapse is tentatively defined as smoking 5 cigarettes in 3 consecutive days since joining the RCT among the 3 study arms.

DETAILED DESCRIPTION:
This research project consists of two parts: (1) Formative study on the use of social networking services for relapse prevention; and (2) A RCT to test the effectiveness of social networking services for relapse prevention 7.1 Phase 1 - Formative study 7.1.1 Study design and objectives Literature review and exploratory data analysis on the existing dataset of ICSCs will be conducted to better define smoking relapse and estimate the relapse rate in the natural setting. In addition, an extensive review of the effectiveness of other similar or relevant intervention studies, including our previous studies and preliminary results of using short messaging services at HKU will be conducted. A consultation group formed by the ICSCs and smoking cessation research team of HKU will be responsible to develop the intervention package through the social networking service, including the content of delivered messages, channels, format, time to be sent, intensity, moderator's protocol, manpower and other logistic arrangement. This intervention package will then be tested in some cognitive interview to assess the relevance, appropriateness, potential effectiveness and acceptance level of the SMS.

7.1.2 Selection of subjects We will invite about 6 quitters (without relapsing for at least one month) and 6 relapsers (smoke 5 cigarettes for 3 days after quitting) from the ICSCs by (i) gender (M, F) and (ii) age group (18-39, 40-59, 60+) to comment on the relevance, appropriateness, potential effectiveness and acceptance level of the intervention package.

7.1.3 Procedures for the cognitive interview The sites for conducting the cognitive interview of the intervention package contents will be the eight ICSCs. A face-to-face semi-qualitative interview will be conducted.

7.1.4 Instruments A semi-structured interview guide and instrument will be used to collect their opinions.

7.1.5 Sample size 12 participants (6 quitters and 6 relapsers) will be recruited. Phase 2 - Randomized controlled trial

1. Study design and objectives: This is a randomized controlled trial (RCT) to compare the relapse rate at the end of the first and third month between participants who join the social network (group A) and those who do not (group B). Research hypothesis: The relapse rate at 1-month and 3-month of the intervention arm (Group A) is lower than the control arm (Group B)
2. Target subjects

   Inclusion criteria:
   * Clients who have received the community-based smoking cessation counseling provided by ICSC
   * Reported tobacco abstinence in the past 7 days at the 8-week follow-up from the first enrollment
   * Aged 18 or above
   * Able to communicate in Cantonese and read Chinese
   * Have a local network mobile phone with mobile internet access

   Exclusion criteria:
   * Those with unstable physical or psychological conditions as advised by the doctor or counselor in charge
   * Smokers with diagnosed alcohol dependence or the score of the Alcohol Use Disorders Identification Test (AUDIT) is 8 or higher
   * Smokers who have difficulties (either physical or cognitive condition) to communicate
   * Currently participating in other smoking cessation programs
3. Procedures:

Smokers who finished the 8-week treatment by TWGHs will be followed up by the staff of TWGHs through telephone or face-to-face visit. Those who meet the inclusion criteria will be introduced the RCT and invited to consent the participation of the RCT through oral or written consent. The social networking service for the intervention group will be available within 3 to 4 days after randomization.

Group A: Intervention arm with relapse prevention intervention in the social group via the social networking service (Potential channel: Whatsapp or Facebook). In order to sustain the abstinence among the participants in the social groups, the intervention content is about how to prevent smoking lapse and relapse, how to deal with high-risk situations and facilitate mutual support among participants. Moderators of the social groups will send messages of brief advice, give feedback to participants' enquiries and facilitate conversations in the platform. We propose the moderator to spend about 1 to 2 hours a day for the social group conversation in a flexible time schedule, and the duration will be at least one month. More details about the intervention will be confirmed at the preparation stage.

Group B: Control arm without any other interventions Counselors, from ICSCs and HKU, who have experience in smoking cessation and familiar with the operation of the social networking service, will be recruited as moderators of the social media groups to deliver the social networking services.

1- and 3-month follow up (after the random allocation) will be conducted by a trained interviewer (blinded to the group assignment) via telephone interview. Subjects who have reported abstinence from smoking at the follow-up will undergo a non-biochemical validation to validate their quitting status. They will be enquired a few questions about their quitting experience and impression, and their family members will be invited to report the smokers' smoking and quitting status thru telephone interview. Also, they will be invited by the interviewer to have biochemical validation tests (saliva cotinine test and exhaled CO test).

4 Randomization and Blinding: Simple randomization method by sequentially numbered, opaque sealed envelopes (SNOSE) will be conducted to ensure both the TWGHs counselors and the participants are masked from the allocation. The counselors who are responsible for the subject recruitment will be masked from the randomization. For each participant who is eligible for the study checked by the counselors, the counselor will call the site randomizer to allocate group identity for the participant by opening one sealed envelope according to the serial number sequentially and inform the counselor for further intervention. Assessors in the follow-ups will not be involved in the randomization process and be totally blinded to the group assignment (single blindness).

5 Instruments: The required baseline information related to demographics and background information will be confirmed at the preparation stage. ICSCs will collect these information from the smokers during the enrollment of the first visit. A structured questionnaire at 1- and 3- month from enrollment of ICSCs will be developed by adopting or modifying international and/or locally validated instruments. The questionnaire gathers information including smoking and quitting history, satisfaction and perceived-usefulness of the social networking services, risk perceptions of smoking, intention to quit smoking (stage of readiness to quit), antecedent factors of the Theory of Planned Behavior model (behavioural beliefs, outcome evaluations, normative beliefs, motivation to comply), pros and cons of smoking (decisional balance), self-efficacy to resist smoking, other lifestyle risk factors (drinking and physical activities), demographic information such as age, gender, marital status, education level and employment status.

6 Sample size determination: Since this is a pilot study to test the feasibility and generate preliminary estimates of effectiveness of the interactive messaging service for smoking cessation, the sample size would be 50 for each arm (i.e. total sample size = 100). Taking reference from the relapse rate (based on the 7-day point prevalence) of ICSCs of TWGH from 2009-2010, 251 out of the 763 quitters at 8 weeks reported that they smoked again at 6 months. In other words, the relapse rate (number of continuing smoking at 6 months among self-reported quitters at the 8-week follow-up) was 33%, assuming no new quitters. We assumed a similar result would occur for the control group of this RCT of relapse prevention (Group B). The effect size is set conservatively at 1:1.5 for the contrast between group A and B. In other words, the estimated relapse rates for A and B are 22% and 33%, respectively. As we only have 100 subjects in total, the power for detecting this difference using the Fisher's exact test is 26%, given alpha is 0.05. That means the study has low probability to reject the alternative hypothesis if it is false. The power would reach to 51.4% when the estimated effect size is set at 1:2. Alternatively, if the total sample size can be increased to 500, the power can reach to 85% for the 1.5 effect size.

7 Methods of statistical analysis Data will be entered into SPSS for Windows (version 20). Descriptive statistics such as frequency, percentage, and mean will be used to summarize the outcomes and other variables. Chi-square tests and t-tests will be used to compare outcome variables between subgroups. Fisher's exact test will be used to compare the quit rates between group A and group B. The intention-to-treat (ITT) analysis will be used such that those lost to contact and refused cases at the follow-ups will be treated as failure to achieve any cessation outcome.

8 Process evaluation To understand the perception and effectiveness of the social networking services, all the participants in the intervention group will also be invited to give feedback through the social networking platform. Furthermore, six participants from the intervention group will be selected (3 relapsers and 3 non-relapsers) to participate in an in-depth interview after the 3-month follow-up. Questions such as their satisfaction, perceptions on the advantages and disadvantages of the intervention, and any other suggestions for improvement will be explored and discussed.

ELIGIBILITY:
Inclusion Criteria:

* Smoked at least 1 cigarette a day when first joined ICSC
* Aged 18 or above at the baseline of the RCT
* Clients who have received 3 to 5 smoking cessation counseling provided by ICSC
* Reported tobacco abstinence in the past 7 days at the 8-week follow-up since receiving treatment from ICSC
* Able to communicate in Cantonese and read Chinese
* Have a local network mobile phone with mobile internet access

Exclusion Criteria:

* Those with unstable physical or psychological conditions as advised by the doctor or counselor in charge
* Smokers with diagnosed alcohol dependence by clinicians or the score of the Alcohol Use Disorders Identification Test (AUDIT) is 8 or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tai Hing Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Integrated Centres on Smoking Cessation (ICSC), Tung Wah Groups of Hospital (TWGH), Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheung YT, Chan CH, Lai CK, Chan WF, Wang MP, Li HC, Chan SS, Lam TH. Using WhatsApp and Facebook Online Social Groups for Smoking Relapse Prevention for Recent Quitters: A Pilot Pragmatic Cluster Randomized Controlled Trial. J Med Internet Res. 2015 Oct 22;17(10):e238. doi: 10.2196/jmir.4829. PMID 26494159

RESULTS

PARTICIPANT FLOW:
Groups:
- WhatsApp: Peer to peer support and delivery of information through WhatsApp for 8 weeks
  Peer to peer support and delivery of information through WhatsApp groups: Intervention arm with relapse prevention intervention in the social group via the social networking service WhatsApp. In order to sustain the abstinence among the participants in the social groups, the intervention content is about (1) Encourage to maintain abstinence; (2) Importance of remaining abstinence; (3) Prevent smoking triggers; (4) Withdrawal symptoms & lapse; (5) Stress and mood management; (6) weight control. We propose the moderator to spend about 1 to 2 hours a day in total for the social group conversation in a flexible time schedule, and the duration of the intervention will be 8 weeks.
- Facebook: Peer to peer support and delivery of information through facebook for 8 weeks
  Peer to peer support and delivery of information through Facebook: Another intervention arm with the same intervention content, but the platform for the participants to share and receive quitting advice is Facebook. They will be strongly suggested to follow the regulations and set up instructions for the participation to protect their privacy.
- Control: No intervention
Period: Overall Study
Arm/Group | WhatsApp | Facebook | Control
Started | 42 | 40 | 54
Completed | 42 | 40 | 54
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Facebook: Peer to peer support and delivery of information through facebook for 8 weeks.
  Peer to peer support and delivery of information through Facebook: Another intervention arm with the same intervention content, but the platform for the participants to share and receive quitting advice is Facebook. They will be strongly suggested to follow the regulations and set up instructions for the participation to protect their privacy.
- Total: Total of all reporting groups
Arm/Group | WhatsApp | Facebook | Control | Total
Number analyzed (Participants) | 42 | 40 | 54 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (10.4) | 37.6 (8.0) | 42.7 (10.4) | 40.5 (9.9)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 11 | 11 | 32
  Male | 32 | 29 | 43 | 104
Region of Enrollment [Number; unit: participants]
  China | 42 | 40 | 54 | 136

OUTCOME MEASURES:

1. Primary Outcome: Self Reported Relapse Rate at 2 Months
Description: Relapse is defined as smoking 5 cigarettes in 3 consecutive days since the most recent quitting. A questionnaire asking smoking status, quitting experience and difficulty in quitting was designed to assess the self reported relapse rate at 2 months.
Time Frame: 2 months after joining the groups for the social networking services.
Measure: Number; unit: participants
Arm/Group | WhatsApp | Facebook | Control
Number analyzed (Participants) | 42 | 40 | 54
participants | 3 | 10 | 13
Statistical Analysis 1: Comparison: WhatsApp vs Control; Test type: Superiority or Other; p = 0.033, Regression, Logistic; Odds Ratio (OR) = 0.21, 95% CI 2-sided [0.05 to 0.89]
Statistical Analysis 2: Comparison: Facebook vs Control; Test type: Superiority or Other; p = 0.934, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.36 to 3.01]

2. Secondary Outcome: Point Prevalence of Self Reported Abstinence for the Previous 7 Days at 2 Months
Description: The outcome was assessed by any self-reported cigarette consumption in the past 7 days at the time of the follow-up. A questionnaire asking smoking status, quitting experience and difficulty in quitting was designed to assess the self reported abstinence for the previous 7 days at 2 months.
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | WhatsApp | Facebook | Control
Number analyzed (Participants) | 42 | 40 | 54
participants | 36 | 28 | 30
Statistical Analysis 1: Comparison: WhatsApp vs Control; Test type: Superiority or Other; p = 0.002, Fisher Exact
Statistical Analysis 2: Comparison: Facebook vs Control; Test type: Superiority or Other; p = 0.199, Fisher Exact

3. Primary Outcome: Self Reported Relapse Rate at 6 Months
Description: Relapse is defined as smoking 5 cigarettes in 3 consecutive days since the most recent quitting. A questionnaire asking smoking status, quitting experience and difficulty in quitting was designed to assess the self reported relapse rate at 6 months.
Time Frame: 6-months
Measure: Number; unit: participants
Arm/Group | WhatsApp | Facebook | Control
Number analyzed (Participants) | 42 | 40 | 54
participants | 11 | 13 | 20
Statistical Analysis 1: Comparison: WhatsApp vs Control; Test type: Superiority or Other; p = 0.285, Regression, Logistic; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.25 to 1.50]
Statistical Analysis 2: Comparison: Facebook vs Control; Test type: Superiority or Other; p = 0.597, Regression, Logistic; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.31 to 1.97]

4. Secondary Outcome: Point Prevalence of Self Reported Abstinence for the Previous 7 Days at 6 Months
Description: The outcome was assessed by any self-reported cigarette consumption in the past 7 days at the time of the follow-up. A questionnaire asking smoking status, quitting experience and difficulty in quitting was designed to assess the self reported abstinence for the previous 7 days at 6 months.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | WhatsApp | Facebook | Control
Number analyzed (Participants) | 42 | 40 | 54
participants | 27 | 19 | 21
Statistical Analysis 1: Comparison: WhatsApp vs Control; Test type: Superiority or Other; p = 0.023, Fisher Exact
Statistical Analysis 2: Comparison: Facebook vs Control; Test type: Superiority or Other; p = 0.527, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | WhatsApp | Facebook | Control
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40 | 0/54
Other Adverse Events (participants affected / at risk) | 0/42 | 0/40 | 0/54

LIMITATIONS AND CAVEATS:
Most subjects had already quit for a few weeks before joining the RCT, so the present RCT did not examine if the intervention helped subjects manage smoking urges at the early stage of quitting. Also, the pilot RCT had small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes